CLINICAL TRIAL: NCT06821490
Title: It is Possible to Reduce the Performance of Axillary Lymphadenectomies in Patients with HER2-positive Breast Cancer with a Clinically Positive Axilla At Diagnosis
Brief Title: Validation of TAD in HER-2 with More Than 2 Lymph Nodes
Acronym: DAD-HER2
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Elvira Buch, Clinical Head of the General Surgery Department, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: DAD-HER2
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Carcinoma Metastatic in Lymph Node; HER2 Positive Breast Carcinoma
Keywords: Targeted Axillary Dissection; HER2-positive breast cance; Two or more diseased axillary lymph nodes at diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- her2positive: Patients who, at diagnosis, have more than 2 affected axillary lymph nodes. Patients in whom the most caudal affected lymph node is marked. After neoadjuvant treatment, a good axillary response is evidenced by ultrasound
  Interventions: Procedure: Targeted axillary dissection and subsequently a lymphadenectomy

INTERVENTIONS:
Procedure: Targeted axillary dissection and subsequently a lymphadenectomy — Selective sentinel lymph node biopsy is performed, along with biopsy of the node marked at diagnosis. Subsequently, a lymphadenectomy is performed, with the three samples separated for pathological study during the same surgical procedure

SUMMARY:
The main objective of the study is to validate the DAT technique in patients with Her2-positive breast cancer who have more than two positive axillary lymph nodes at diagnosis. After receiving adequate oncological treatment and axillary assessment by ultrasound for complete radiological response, DAT and Berg level I and II lymphadenectomy will be performed to assess false negatives and positives, as well as their sensitivity and specificity.

DETAILED DESCRIPTION:
This study aims to determine whether axillary treatment can be further de-escalated in patients with HER2-positive breast cancer, as this group has shown good responses to certain targeted therapies. It focuses on reducing the need for extensive axillary surgery (known as axillary lymphadenectomy or AL), which can cause complications, by using a less invasive procedure called Targeted Axillary Dissection (TAD). This method combines the removal of sentinel lymph nodes and previously marked nodes, allowing for an assessment of treatment response without needing to remove all lymph nodes. Currently, this method is used in patients diagnosed with axillary disease involving fewer than two axillary nodes.

Main Objective:

To evaluate whether axillary lymphadenectomy can be avoided in HER2-positive breast cancer patients with more than two affected axillary nodes who respond well to chemotherapy before surgery.

Secondary Objectives:

Analyze the oncological treatment response in these patients. Determine how many affected nodes respond to the treatment. Evaluate whether the number of affected nodes at diagnosis limits the possibility of performing TAD.

Compare methods for locating the affected nodes. Verify the concordance between marked nodes and sentinel nodes.

Methodology:

This is a multicenter, prospective descriptive study. Women with HER2-positive breast cancer who receive chemotherapy before surgery will be included. Those who show a good axillary response will be offered the TAD procedure, followed by lymphadenectomy, to assess the sensitivity, specificity, false negatives, and true positives of the technique. Clinical and radiological data will be collected to analyze outcomes and complications.

Significance:

The TAD procedure has already allowed this hospital to reduce extensive axillary surgeries by 30%, preventing associated complications. This study seeks to confirm whether this approach is safe and effective in a specific group of HER2-positive breast cancer patients with more than two affected nodes at diagnosis. If successful, it could lead to a change in how these patients are treated, reducing risks and improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1 (physical condition: able to walk and live a normal life)
* Patients with early-stage breast cancer (BC) with histopathological diagnosis of HER2+ and axillary involvement.

Patients with either positive or negative hormonal receptor expression will be included.

* Patients must have marked the pathological axillary lymph node.
* Any number of affected or suspicious lymph nodes at diagnosis is allowed.
* Patients will receive appropriate neoadjuvant treatment based on a combination of chemotherapy and anti-HER2 therapy.

  • After neoadjuvant treatment and prior to surgery, radiological response will be assessed.
* No relevant comorbidities, adequate liver and kidney function, and no contraindications to receive neoadjuvant treatment followed by surgery and radiotherapy.

Exclusion Criteria:

* Patients with inoperable breast cancer.
* Patients with a diagnosis of inflammatory breast cancer.
* Patients without a diagnostic biopsy of the suspicious lymph node or the presence of axillary conglomerate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with HER2+ breast cancer, with more than two affected lymph nodes at diagnosis, who receive chemotherapy. These patients have been marked at diagnosis and show a good response after neoadjuvant treatment
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Location of the marked lymph node and the sentinel lymph node, and assessment after lymphadenectomy of number of true positives and negatives, sensitivity and specificity | From enrollment to the end of treatment at 12 months
  Determining the number of positive and negative nodes in targeted axillary dissection and axillary lymphadenectomy

SECONDARY OUTCOMES:
Detection of the axillary lymph node marked at diagnosis and Detection of the sentinel lymph node and concordance between marked lymph node and sentinel lymph node | From enrollment to the end of treatment at 12 months
  Number of marked nodes that match the sentinel nodes
Number of positive lymph nodes at diagnosis | From enrollment to the end of treatment at 12 months
  Number of positive lymph nodes at the time of diagnosis for which TAD (directed axillary

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico de la Comunidad Valenciana, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data will be protected in the patient's medical record, although the patient is informed about the study and will sign a consent form. It is uncertain whether it is ethical to share the individual data.

REFERENCES:
- [Background] Ng S, Sabel MS, Hughes TM, Chang AE, Dossett LA, Jeruss JS. Impact of Breast Cancer Pretreatment Nodal Burden and Disease Subtype on Axillary Surgical Management. J Surg Res. 2021 May;261:67-73. doi: 10.1016/j.jss.2020.12.007. Epub 2021 Jan 6. PMID 33421795
- [Background] Gasparri ML, de Boniface J, Poortmans P, Gentilini OD, Kaidar-Person O, Banys-Paluchowski M, Di Micco R, Niinikoski L, Murawa D, Bonci EA, Pasca A, Rubio IT, Karadeniz Cakmak G, Kontos M, Kuhn T. Axillary surgery after neoadjuvant therapy in initially node-positive breast cancer: international EUBREAST survey. Br J Surg. 2022 Aug 16;109(9):857-863. doi: 10.1093/bjs/znac217. PMID 35766257
- [Background] Simons JM, Jacobs JG, Roijers JP, Beek MA, Boonman-de Winter LJM, Rijken AM, Gobardhan PD, Wijsman JH, Tetteroo E, Heijns JB, Yick CY, Luiten EJT. Disease-free and overall survival after neoadjuvant chemotherapy in breast cancer: breast-conserving surgery compared to mastectomy in a large single-centre cohort study. Breast Cancer Res Treat. 2021 Jan;185(2):441-451. doi: 10.1007/s10549-020-05966-y. Epub 2020 Oct 19. PMID 33073303
- [Background] Galimberti V, Ribeiro Fontana SK, Vicini E, Morigi C, Sargenti M, Corso G, Magnoni F, Intra M, Veronesi P. "This house believes that: Sentinel node biopsy alone is better than TAD after NACT for cN+ patients". Breast. 2023 Feb;67:21-25. doi: 10.1016/j.breast.2022.12.010. Epub 2022 Dec 20. PMID 36566690
- [Background] Cha C, Ahn SG, Kim D, Lee J, Park S, Bae SJ, Kim JY, Park HS, Park S, Kim SI, Park BW, Jeong J. Axillary response according to neoadjuvant single or dual human epidermal growth factor receptor 2 (HER2) blockade in clinically node-positive, HER2-positive breast cancer. Int J Cancer. 2021 Oct 15;149(8):1585-1592. doi: 10.1002/ijc.33726. Epub 2021 Jul 8. PMID 34213778
- [Background] Bernet L, Piñero A, Martínez M, Sicart SV, Algara M, Palomares E. Consensus of the Spanish Society of Breast Senology and Pathology (SESPM) on Selective Biopsy of the Sentinel Node (BSGC) and axylar management in breast cancer (2022). Revista de Senologia y Patologia Mamaria. 2022 Oct 1;35(4):243-59.
- [Background] Early Breast Cancer Trialists' Collaborative group (EBCTCG). Trastuzumab for early-stage, HER2-positive breast cancer: a meta-analysis of 13 864 women in seven randomised trials. Lancet Oncol. 2021 Aug;22(8):1139-1150. doi: 10.1016/S1470-2045(21)00288-6. PMID 34339645
- [Background] Schettini F, Pascual T, Conte B, Chic N, Braso-Maristany F, Galvan P, Martinez O, Adamo B, Vidal M, Munoz M, Fernandez-Martinez A, Rognoni C, Griguolo G, Guarneri V, Conte PF, Locci M, Brase JC, Gonzalez-Farre B, Villagrasa P, De Placido S, Schiff R, Veeraraghavan J, Rimawi MF, Osborne CK, Pernas S, Perou CM, Carey LA, Prat A. HER2-enriched subtype and pathological complete response in HER2-positive breast cancer: A systematic review and meta-analysis. Cancer Treat Rev. 2020 Mar;84:101965. doi: 10.1016/j.ctrv.2020.101965. Epub 2020 Jan 17. PMID 32000054
- [Background] Haque W, Verma V, Hatch S, Suzanne Klimberg V, Brian Butler E, Teh BS. Response rates and pathologic complete response by breast cancer molecular subtype following neoadjuvant chemotherapy. Breast Cancer Res Treat. 2018 Aug;170(3):559-567. doi: 10.1007/s10549-018-4801-3. Epub 2018 Apr 24. PMID 29693228